CLINICAL TRIAL: NCT03042507
Title: Psychosocial Intervention for Young Children With Chronic Tics
Acronym: CBIT JR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of California, Los Angeles (Other); University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012011424R005
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Tourette's Syndrome; Tourette's Disorder; Tourette's Disease; Tourette Disorder; Tourette Disease; Tic Disorder, Combined Vocal and Multiple Motor; Multiple Motor and Vocal Tic Disorder, Combined; Gilles de La Tourette's Disease; Gilles de la Tourette Syndrome; Gilles De La Tourette's Syndrome; Combined Vocal and Multiple Motor Tic Disorder; Combined Multiple Motor and Vocal Tic Disorder; Chronic Motor and Vocal Tic Disorder
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Trial (Other): This is a non-randomized open trial of a behavioral intervention for young children with tics
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT)

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT) — The existing CBIT protocol includes a functional assessment procedure designed to identify relevant contextual variables (both antecedent and consequent) impacting tic expression and guide the development of an individualized behavioral program to neutralize these contextual influences in the service of tic reduction and psychoeducational component. Given the central role that negative social reactions typically play in tic exacerbation and maintenance, psychoeducation about tics is systematically provided to parents, siblings, and other caretakers and prominent individuals in the child's life. The other primary CBIT component, Habit Reversal Training (HRT), is used to weaken or eliminate the negative reinforcement cycle created by tic-contingent reduction in premonitory urge.

SUMMARY:
Analysis of data from the recently completed NIH Child Comprehensive Behavioral Intervention for Tics (CBIT) study found a manualized behavioral treatment approach strongly superior to psychoeducation/supportive therapy for reducing tic severity in 9-16 year-old youths with TS or other Chronic Tic Disorders. Buoyed by the success of the NIH study, the research group now seeks to extend and disseminate the CBIT treatment through the systematic adaptation of the CBIT protocol for use across a broader range of ages and treatment settings.

The goal of the this project is to develop a downward extension of the CBIT therapist guide and parent workbook for use in 4-8 year old children with chronic tics. The revised CBIT-JR manual/workbook will be pilot tested in five children at each of the three study sites (UCLA, UWM, Weill Cornell) in order to provide initial data regarding treatment feasibility and acceptability as well as our ability to implement the new intervention, along with relevant quality control procedures, consistently across sites. These pilot data will then be used to seek R01 support for a larger controlled multisite trial examining the efficacy of CBIT-JR.

Although arguably more complex than a single-site design, we have opted for a multsite study in order: 1) to take advantage of the established productive collaborative relationship and collective expertise in childhood tic disorders and psychosocial treatment development across our three sites, 2) to collect the proposed feasibility data in a much shorter period of time than otherwise possible, and as noted above 3) to demonstrate the cross-site portability of the treatment - which will be necessary if we are to obtain subsequent funding for a larger-scale efficacy trial.

DETAILED DESCRIPTION:
The overall aim of the proposed project is to develop and obtain preliminary feasibility and acceptability data for a family-based behavioral intervention to reduce tic severity and the negative impact of TS-related symptoms in young children (ages 4-8) with chronic tics and Tourette syndrome. This intervention entails the use of targeted psychoeducation about tics and related conditions and a functional analytic protocol designed to identify and correct environmental influences thought to exacerbate and/or maintain child tic expression. Although similar to the family-based component used in our recently completed CBITS trial for older children, an independent body of literature supports the efficacy of functional analysis for ameliorating a variety of both behaviorally and biologically-driven behaviors. The investigators will work with an early child interventionist to adapt the current family-based protocol for younger children. The new manual will then be feasibility tested in anticipation of a larger externally-funded trial to further develop and evaluate the efficacy of this intervention.

More specifically, the study aims are to:

1. Adapt the current CBIT Manual for use with the families of 4-8 year old children with chronic tic disorder. Our revision will be informed by a meeting of the study PI's and Dr. Mary O'Connor, an early childhood interventionist at UCLA to review our current family-intervention and other treatment protocols targeting related psychopathology in young children.
2. Document the feasibility, acceptability, and cross-site portability of the new manual in a small open trial of 15 youngsters (five each at UCLA, UWM, and Weill Cornell).

ELIGIBILITY:
Inclusion Criteria:

1. age 4-8
2. presence of motor and/or vocal tics for at least 6 months.
3. tics are of at least moderate clinical severity as evidenced by a Clinical Global Impressions (CGI) Severity score of 4 or higher (tic symptoms clearly noticeable to family and occasionally to families and associated with at least some minimal level of distress and/or interference.
4. free of PDD or other developmental disability
5. IQ estimate of 70 or higher
6. comorbid disorder (e.g., ADHD, OCD, ODD) will be allowed provided that the tic symptoms are of primary concern to parents and comorbid symptoms are not of sufficient severity to require immediate treatment other than that provided by the current study.
7. pre-existing stable medication, tic or otherwise, will also be allowed provided the family agrees to refrain from med changes over the course of the study if at all possible.
8. sufficient command of the English language to comply with study protocol.

Exclusion Criteria:

-

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2012-01-20 (Actual); Primary Completion 2012-12-29 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS). | Baseline, week 8
  Change in tic severity from baseline to week 8 as measured by the YGTSS.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bennett, PhD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: Yes